CLINICAL TRIAL: NCT00760162
Title: Pilot-Scale Clinical Trials of Kibow Biotics® (a Patented and Proprietary Probiotic Formulation) in Chronic Kidney Failure
Brief Title: Pilot-Scale Clinical Trials of Kibow Biotics® in Chronic Kidney Failure
Acronym: Probiotics
Status: Completed | Type: Observational
Sponsor: Kibow Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: KIB001
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Chronic Kidney Failure
Keywords: Chronic Kidney failure stage three and four; Probiotics; Kibow Biotics; Enteric Dialysis; Gut based removal uremic toxin removal
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- HSCB, Brooklyn, NY: State University of New York Brooklyn, NY 11203
- 2. Nephrology Associates,: Scarborough, ON CANADA, LI H IC5
- 3.New York Harbor VA Medical Center: NYU School of Medicine New York, NY.10010
- 4.Hospital Juarez De Mexico: Madero, Mexico, D.FC.P. 07760
- 5. Hospital Italiano de Buenos Aires: Buenos Aires, Argentina.
- 6. National Hospital: Abuja, Nigeria

SUMMARY:
The bowel can serve as a complement to the kidneys' excretory function

A specifically formulated probiotic product comprised of defined and tested microbial strains may afford renoprotection in what has been called "enteric dialysis"® Confirm the alleviation of uremic syndrome hypothesis Determine the outcome of probiotics treatment Confirm U.S. FDA's Generally Recognized As Safe (GRAS) status - if needed

DETAILED DESCRIPTION:
Probiotics are increasingly utilized clinically. As their safety and health benefits are established, it is reasonable to anticipate that probiotic bacteria will be incorporated into a growing number of clinical regimens.

Following exploratory testing of orally administered probiotic bacteria in rats and minipigs with surgically induced chronic kidney disease (CKD), a trial is now in progress to determine whether daily treatment with gastrointestinal (GI) probiotic bacteria will delay the onset of and/or improve established signs and symptoms of human CKD.

To assess the potential benefit in devising a gut-based probiotic formulation (Kibow Biotics®) as a dieatary supplement - Over The Counter (OTC)product in CKD applications.

Extensive in vitro R&D investigations in Kibow's laboratories

Simulated Human Intestinal Microbial Ecosystem (SHIME, Ghent University, Belgium) utilized in a computer-controlled in vitro system validated the concept that the chosen microbial formulation would metabolize and reduce concentration of nitrogenous components including urea, creatinine, and uric acid. Bacterial strains studied were Streptococcus thermophilus (KB27), Lactobacillus acidophilus (KB31) and Bifidobacterium longum (KB35).

Oral administration of these bacterial formulations, tested in the 5/6th nephrectomized rat model (at Thomas Jefferson University, Phila., PA) and minipig model (at Indiana University, Indianapolis, IN), decreased both blood urea nitrogen (BUN) and serum creatinine (Scr) levels.

Two independent veterinarians investigated the effect of Kibow Biotics® on clinically manifested renal failure in uremic cats and dogs of both genders and varying body weights. Based on positive results, this formulation, marketed and distributed as AzodylTM, is currently licensed for veterinary applications to Vetoquinol USA

ELIGIBILITY:
Inclusion Criteria:

* CKD patients Stage III and IV
* 18 to 75 years old, able and willing to give an informed consent
* Baseline serum creatinine > 2.5 mg/dL

Exclusion Criteria:

* Women who are pregnant or nursing
* Patients who are on antibiotic treatment at the time of screening will be excluded from the study (Patients who have received antibiotics should have stopped them for at least 14 days prior to screening)
* Patients who do not agree to sign the informed consent form
* Active dependency on drugs or alcohol
* Patients with documented Human Immunodeficiency Virus (HIV) infection/ Acquired Immunodeficiency Syndrome (AIDS)/Liver Disease
* Any medical, psychiatric, debilitating disease/disorder or social condition that in the judgment of the investigator would interfere with or serve as a contraindication to adherence to the study protocol or ability to give informed consent, or affect the overall prognosis of the patient
* Patients who are on coumadin therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Out patient Hospital setting
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2007-08; Primary Completion 2009-07 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
PRIMARY: Changes in blood chemistry - BUN, Creatinine and Uric acid | six months
Changes in BUN, Creatinine and uric acid levels | six months

CONTACTS AND LOCATIONS:
Overall Officials: Eli A Friedman, MD, Study Chair — Downstate Medical Center - State University of New York, Brooklyn, NY
Locations (2):
- United States (2):
  - Downstate Medical Center,HSCB, State University of New York, Brooklyn, New York
  - SUNY DownState Medical Center-Renakl Division, Brooklyn, New York

REFERENCES:
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148
- [Derived] Ranganathan N, Friedman EA, Tam P, Rao V, Ranganathan P, Dheer R. Probiotic dietary supplementation in patients with stage 3 and 4 chronic kidney disease: a 6-month pilot scale trial in Canada. Curr Med Res Opin. 2009 Aug;25(8):1919-30. doi: 10.1185/03007990903069249. PMID 19558344